CLINICAL TRIAL: NCT00191126
Title: Randomized Phase III Trial of Surgery Alone or Surgery Plus Preoperative Gemcitabine-Cisplatin in Clinical Early Stages(T2N0, T1 - 2N1, T3N0 AND T3N1) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Randomized Phase III Trial of Surgery Alone or Surgery Plus Preoperative Gemcitabine-Cisplatin in Early Stages NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3532; B9E-MC-S132 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other)
  Interventions: Procedure: surgery
- B (Experimental)
  Interventions: Drug: gemcitabine; Drug: Cisplatin; Procedure: surgery

INTERVENTIONS:
Drug: gemcitabine — 1250 mg/m2, IV, day 1 and 8, q 21 days x 3 cycles
  Other Names: LY188011; Gemzar
  Arms: B
Drug: Cisplatin — 75 mg/m2, IV, q 21 days x 3 cycles
  Arms: B
Procedure: surgery — surgery

SUMMARY:
Preoperative chemotherapy is considered to play a role in early stage non small cell lung cancer (NSCLC) .The use of preoperative Cisplatin/Gemcitabine chemotherapy has proven feasible and without excessive morbidity or mortality in the Phase II setting. The aim of the present Phase III study is to determine whether 3 cycles of preoperative chemotherapy with Cisplatin/Gemcitabine improves progression free survival of NSCLC patients versus surgery alone. Postoperative chemotherapy will not be utilized in this Phase III trial.

ELIGIBILITY:
Main inclusion Criteria:

* Must have pathologic documentation of non-small cell lung cancer, IB, II, IIIA.
* ECOG Performance Status of 0 - 1
* Bidimensionally measurable disease or evaluable disease
* Adequate organ function

Main exclusion Criteria:

* Have greater than Grade 1 neuropathy - motor/sensory
* Significant history of cardiac disease
* Pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2000-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | baseline to measure progressive disease

SECONDARY OUTCOMES:
To compare the survival and sites of relapse in the two study arms. | baseline to progressive disease
Pharmacology toxicity | every cycle
Response rate | baseline to measured progressive disease
Pathologic response rate of tissue samples | baseline, post chemotherapy, post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (37):
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Liège
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Sarajevo, Bosnia and Herzegovina
- Bulgaria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Varna
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Cairo, Egypt
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Tallinn, Estonia
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Löwenstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Ulm
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Pécs, Hungary
- Italy (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Chieti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., L’Aquila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Siena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Teramo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Verona
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Klaipedos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Vilnius
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Warsaw, Poland
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Cluj-Napoca
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Riyadh, Saudi Arabia
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Košice
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Helsingborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Malmo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician., Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Scagliotti GV, Pastorino U, Vansteenkiste JF, Spaggiari L, Facciolo F, Orlowski TM, Maiorino L, Hetzel M, Leschinger M, Visseren-Grul C, Torri V. Randomized phase III study of surgery alone or surgery plus preoperative cisplatin and gemcitabine in stages IB to IIIA non-small-cell lung cancer. J Clin Oncol. 2012 Jan 10;30(2):172-8. doi: 10.1200/JCO.2010.33.7089. Epub 2011 Nov 28. PMID 22124104
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com